CLINICAL TRIAL: NCT02010983
Title: Screening for Dysplasia in Longstanding Idiopathic Achalasia: a Prospective Study
Brief Title: Achalasia and Dysplasia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Guy Boeckxstaens, Prof. Dr., KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S55021
Record Dates: First submitted 2013-02-14; First posted 2013-12-13 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Dysplasia in Longstanding Achalasia; Relation Between Food Stasis and Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- longstanding achalasia (Experimental)
  Interventions: Other: chromoendoscopy

INTERVENTIONS:
Other: chromoendoscopy — chromoendoscopy (lugol stain and virtual chromoendoscopy)

SUMMARY:
Patient with achalasia have a 10-50 fold increased risk to develop esophageal squamous cell carcinoma (ESCC). Early diagnosis of ESCC is essential, and detection of an earlier dysplastic stage is preferred. Endoscopic detection is however difficult and often delayed. Chromoendoscopy with Lugol dye increases detection rates dysplasia and ESCC to 91-100%. The aim of this study was therefore to evaluate a screening program using chromoendoscopy with Lugol to detect dysplasia in patients with idiopathic achalasia.

A second objective is to study the relationship between foodstasis and the development op dysplasia

ELIGIBILITY:
Inclusion Criteria:

* longstanding achalasia (> 15y)
* > 18y old
* informed consent

Exclusion Criteria:

* allergy to iodine
* esophageal carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-10; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
incidence of dysplasia in patients with longstanding achalasia | 1 year

SECONDARY OUTCOMES:
additive value of chromoendoscopy in comparison with lugol stain | 1 year
relationship between food stasis and dysplasia | 1 year
  * relationship between elevated LES pressure and dysplasia
  * relationship between stasis on EndoFLIP and dysplasia
  * relationship between stasis on timed barium esophagogram and dysplasia

CONTACTS AND LOCATIONS:
Locations (1):
- UZleuven, Leuven, Belgium